CLINICAL TRIAL: NCT04720976
Title: A Phase 1/2a, Multicenter, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Evidence of Antitumor Activity of JAB-3312 Based Combination Therapies in Adult Patients With Advanced Solid Tumors
Brief Title: JAB-3312 Based Combination Therapy in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JAB-3312-1003
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor; NSCLC
Keywords: KRAS G12C, EGFR
MeSH Terms: interventions — binimetinib; pembrolizumab; sotorasib; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- JAB-3312+Pembrolizumab dose escalation (Experimental): Dose escalation
  Interventions: Drug: JAB-3312; Drug: Pembrolizumab
- JAB-3312+ Binimetinib dose escalation (Experimental): Dose escalation
  Interventions: Drug: JAB-3312; Drug: Binimetinib
- JAB-3312+Pembrolizumab dose expansion (Experimental): Dose expansion
  Interventions: Drug: JAB-3312; Drug: Pembrolizumab
- JAB-3312+Binimetinib dose expansion (Experimental): Dose expansion
  Interventions: Drug: JAB-3312; Drug: Binimetinib
- JAB-3312+Sotorasib dose escalation (Experimental): Dose escalation
  Interventions: Drug: JAB-3312; Drug: Sotorasib
- JAB-3312+ Osimertinib dose escalation (Experimental): Dose escalation
  Interventions: Drug: JAB-3312; Drug: Osimertinib
- JAB-3312+ Sotorasib dose expansion (Experimental): Dose expansion
  Interventions: Drug: JAB-3312; Drug: Sotorasib
- JAB-3312+ Osimertinib dose expansion (Experimental): Dose expansion
  Interventions: Drug: JAB-3312; Drug: Osimertinib

INTERVENTIONS:
Drug: JAB-3312 — JAB-3312 will be administered orally, variable dose.
Drug: Binimetinib — Binimetinib will be administered orally.
  Arms: JAB-3312+ Binimetinib dose escalation; JAB-3312+Binimetinib dose expansion
Drug: Pembrolizumab — Pembrolizumab will be administered as an intravenous infusion.
  Arms: JAB-3312+Pembrolizumab dose escalation; JAB-3312+Pembrolizumab dose expansion
Drug: Sotorasib — Sotorasib will be administered orally.
  Arms: JAB-3312+ Sotorasib dose expansion; JAB-3312+Sotorasib dose escalation
Drug: Osimertinib — Osimertinib will be administered orally.
  Arms: JAB-3312+ Osimertinib dose escalation; JAB-3312+ Osimertinib dose expansion

SUMMARY:
To evaluate the safety and tolerability of JAB-3312 administered in investigational regimens in adult participants with advanced solid tumors.

DETAILED DESCRIPTION:
To assess the safety and tolerability and determine the Recommended phase 2 dose (RP2D) of JAB-3312 in combination with PD1 inhibitor or MEK inhibitor in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed metastatic or locally advanced solid tumor. Some cohorts must meet specific expression or gene mutation where indicated
* Sufficient organ function
* Participants must have at least 1 measurable lesion as defined by RECIST v1.1
* Must be able to provide an archived tumor sample
* ECOG performance status score of 0 or 1.

Exclusion Criteria:

* History of cancer that is histologically distinct from the cancers under study
* Active or untreated central nervous system (CNS) metastases
* History of pneumonitis or interstitial lung disease (ILD)
* Has active hepatitis B, hepatitis C infection, HIV
* Any severe and/or uncontrolled medical conditions
* LVEF ≤50%
* QTcF >470 msec

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities | 24 months
  Incidence of dose limiting toxicities (DLTs) in the dose escalation phase. A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first treatment cycle. (Dose escalation phase)
Objective response rate (ORR) | 24 months
  ORR is defined as the proportion of participants with complete response or partial response (CR+PR). (Dose expansion phase)
Duration of response (DOR) | 24 months
  DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy, to disease progression or death due to any cause, whichever occurs first. (Dose expansion phase)
Duration of response (DCR) | 24 months
  DCR is defined as proportion of participants with complete response, partial response, stable disease(CR+PR+SD). (Dose expansion phase)
Progression-free survival (PFS) | 24 months
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression or death which occurs first. (Dose expansion phase)
Overall survival (OS) | 24 months
  OS is defined as the interval of time between the date of first treatment until death, loss to follow up or termination of the study by the sponsor. (Dose expansion phase)
Number of participants with adverse events | 24 months
  All patients participating in this study will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs, electrocardiograms, cardiac imaging and ophthalmological assessments (Dose escalation phase)

SECONDARY OUTCOMES:
Objective response rate (ORR) | 24 months
  ORR is defined as the proportion of participants with complete response or partial response (CR+PR). (Dose escalation phase)
Duration of response (DOR) | 24 months
  DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy, to disease progression or death due to any cause, whichever occurs first. (Dose escalation phase)
Duration of response (DCR) | 24 months
  DCR is defined as proportion of participants with complete response, partial response, stable disease(CR+PR+SD). (Dose escalation phase)
Progression-free survival (PFS) | 24 months
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression or death which occurs first. (Dose escalation phase)
Overall survival (OS) | 24 months
  OS is defined as the interval of time between the date of first treatment until death, loss to follow up or termination of the study by the sponsor(Dose escalation phase)
Plasma concentration (Cmax) | 24 months
  Highest observed plasma concentration of JAB-3312(dose escalation phase)
Time to achieve Cmax (Tmax) | 24 months
  Time of highest observed plasma concentration of JAB-3312(dose escalation phase)
Area under the plasma concentration-time curve (AUC) | 24 months
  Area under the plasma concentration time curve of JAB-3312(dose escalation phase)
Number of participants with adverse events | 24 months
  All patients participating in this study will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs, electrocardiograms, cardiac imaging and ophthalmological assessments (Dose expansion phase)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Los Angeles, California
  - Research Site, New Haven, Connecticut
  - Research Site, Jacksonville, Florida
  - Research Site, Orange City, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Detroit, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah

REFERENCES:
- [Derived] Kang D, Wang Y, Lin Y, Ma WW, Morgensztern D, Leventakos K, Bi C, Ding Y, Xiong J, Yan M, Sun X, Wang P, Ma C, Wang Y. JAB-3312, a Potent Allosteric SHP2 Inhibitor That Enhances the Efficacy of RTK/RAS/MAPK and PD-1 Blockade Therapies. Clin Cancer Res. 2025 Jul 15;31(14):3019-3032. doi: 10.1158/1078-0432.CCR-24-3691. PMID 40333694